CLINICAL TRIAL: NCT06076707
Title: Comparing Post-operative Analgesic Effectiveness of Wound Infiltration Using Bupivacaine, Tramadol, and Tramadol Plus Bupivacaine in Patients Undergoing Elective Cesarean Section Under Spinal Anesthesia at Dessie Comprehensive Specialized Hospital, Ethiopia 2022 a Double-Blinded Control Study.
Brief Title: Comparing Analgesic Effects of Wound Infiltration Using Bupivacaine, Tramadol, and Tramadol Plus Bupivacaine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wollo University (Other)
Responsible Party: Principal Investigator, Aynalem Befkadu Woldemichael, Quality control coordinater, Research team leader, lecturer in anesthesia, Wollo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1989156
Record Dates: First submitted 2023-05-17; First posted 2023-10-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The data collector and the investigator will be blind for the study while the patient is not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tramadol (T) group (Experimental): Participants will be infiltrated with only 200mg tramadol around the wound.
  Interventions: Drug: bupivacain-tramadol
- Bupivacain (B) group (Placebo Comparator): participants will be infiltrated with only bupivacaine around the wound
  Interventions: Drug: bupivacain-tramadol
- Tramadol + bupivacain ( T+B) group (Experimental): The participants will be infiltrated with tramadol and bupivacaine which are mixed together in the same syringe.
  Interventions: Drug: bupivacain-tramadol

INTERVENTIONS:
Drug: bupivacain-tramadol — Comparing effectiveness of tramadol and bupivacaine for postoperative pain treatment and prevention for cesarian section

SUMMARY:
The goal of this study's clinical trial is to compare in post-operative analgesic effectiveness of wound infiltration using bupivacaine, tramadol, and tramadol plus bupivacaine in patients undergoing elective cesarean section under spinal anesthesia. The main question the study aimed to answer is "which approach is best among the 3"

all participants need to respond to the pain severity for the data collectors and they will receive treatments accordingly There will be 3 groups in the study

* group T: for tramadol
* group B: for bupivacaine
* group TB : tramadol + bupivacaine

DETAILED DESCRIPTION:
Source Population: All parturients who are scheduled for elective cesarean delivery under spinal anesthesia at Dessie Comprehensive Specialized Hospital

Sample size determination: since there is no previous study done with this title in the study area, we take from a previous study done by Sahmeddini et al in India in the same population. We choose the "time for the first request of analgesia" variable because we found a larger sample size with this variable using the G*Power application. Using G*Power (using version 3.1.9.2) with a power of 80% and confidence interval of 95%, we estimated 153 participants, and considering dropout and nonresponse (10% contingency) a total of 163 patients (54 in each group) would be needed.

Sampling procedure

A 5-month logbook report of the hospital showed that around 400 patients undergo elective c/s. 163 patients will be recruited with a probability of 24% until the sample size is achieved by considering the sequential patients scheduled for C/S as the sampling frame. All patients have a 50% equal chance of being included in the study. The first patient will be recruited by lottery method and then every 2nd will be included until the required sample size is completed. After informed consent is taken, eligible participants will be allocated to one of the two groups with a sealed non-transparent envelope containing the name of the study group

Data collection procedure:

4 anesthetists will be trained by the principal investigator about "how to perform their given tasks" in the research for 5 days. There will be 2 BSC anesthetists dedicated to data collection, 1 BSC anesthetist maintaining randomization and preparing the drugs, and 1 MSC anesthetist performing local infiltration. Explanation about the study and taking written informed consent will be done by the data collectors. The routine peri-operative spinal anesthesia care will be maintained and the interventional drugs will be administered at the end of the procedure before wound closure. The data collector will meet the patient in PACU for the second time and start to assess pain intensity, tramadol consumption, time for the first analgesic request as well as adverse side effects using systematically structured questionnaires and chart review. The supervisors will assist and supervise the data collection process. All data collectors will be BSc anesthetists who have three years of experience. An evaluation will be performed at eight different time points: T0, T2, T4, T6, T8, T12, T18, and T24. Collected data will be checked for completeness, accuracy, and clarity by the principal investigator and the supervisors. For measuring and comparing the intensity and prevalence of pain, NRS has been found to be reliable in a rural population irrespective of literacy status(29)

Blinding

The data collector, patient, and primary investigators will be blinded about the components of drugs in the wound infiltration. The interventional drugs will be prepared by another anesthetist who will not participate in data collection or as an investigator. He/ she will prepare an envelope that will be generated by computer software for all study participants and held sealed until the day of surgery. On the day of surgery after they change clothes the mother will pick up the envelope that will open by one anesthetist who will be responsible for writing the generated random number and letter as TB for tramadol + bupivacaine group and T for tramadol group and B for bupivacaine group.

Data quality management

Training will be given to data collectors regarding study tools, objectives of the study, rights of respondents, and confidentiality of the information. To ensure the quality of data, we will check out for completeness, accuracy, and clarity before data entry. The complete data will enter into the SPSS version 22 computer program. Data clean-up and cross-checking will before analysis.

Data processing and statistical analysis

Data will be checked, coded, entered, and analyzed by SPSS version 22 computer program. The normality of data will be checked by K using the Shapiro-Wilk normality test and homogeneity of variance by Levene's test. The presence of Outliers will also be assessed by a boxplot. Analysis of variance (ANOVA) and Kruskal-Wallis H test will be used for normally distributed continuous data and non-normally distributed or non-parametric data respectively. If these ANOVAs or Kruskal-Wallis H test e significant, then Tukey post hoc test was used to compare one group with the others. Categorical data will be analyzed using the Pearson Chisquared test. Data were expressed as a mean and standard deviation (SD) and Median (Q1-Q3). Frequency, percentages, tables, and figures will be used to summarize data. Data will be expressed in terms of mean ± SD for normally distributed data or median (interquartile range) for skewed data. P-value < 0.05 with a power of 80% is considered statistically significant.

Standard operating procedure (Anesthesia protocol) Step 1: Preparation A standard preoperative assessment will be done for all parturients one day before the surgery. All mothers will receive premedication (dexamethasone 8mg, metoclopramide 10mg, and cimetidine 200mg). All necessary equipment like anesthesia mashie, suction machine, oxygen supply, vaporizers, Pulse oximetry, ECG, BP, Capnography (if applicable), Face mask, Oro pharyngeal airway, ETT, LMA (if appropriate), Boogie or Stylet and the spinal set will be checked and prepared. Availability of inductional, relaxants, antiemetics, analgesia, Local anesthetics, and emergency drugs should be checked before the parturient enters the OR. We may not need all these equipment and drugs for SA but we may face failed spinal, high spinal, or total spinal so we should have a backup plan.

Step 2: SA administration and intra-op SA management After the mother entered the OR and is placed on the OR table, SA will be performed by one BSC anesthetist between L3-L4 interspace at sitting position by using tuffers line as a landmark with a 25 gauge spinal needle and 12.5 ml of 0.5% isobaric bupivacaine at a rate of 0.2 ml per second. Then routine intraoperative SA care will be provided for all parturients.

Step 3: Wound infiltration All interventional drugs will be prepared 10 minutes before the end of surgery in a 10cc syringe. At the end of surgery before wound closure, group T will receive 2 mg/kg tramadol, group B will receive 0.25% of 0.7ml/kg bupivacaine and TB will receive a combination of tramadol (2mg/kg and bupivacaine (0.25%, 0.7ml/kg) as wound site infiltration by MSC anesthetist. Then after checking vital signs, all parturients will transfer to PACU and will meet the data collector for the second time.

Operational definition Wound infiltration: the analgesic technique of administering local anesthetic with or without additives directly into the surgical incision at the end of the procedure.

Acute postoperative pain: is the pain experienced immediately after an operation, usually lasting for days or sometimes weeks Chronic pain: is any pain that remains or keeps coming back for more than 3 months or for longer than the expected healing time.

Chronic post-surgical pain: pain that develops after a surgical procedure that lasts for at least three months.

Postoperative pain: when patients complain about the presence of pain after an operation or any pain score other than zero within 24 hours.

Cesarean delivery: delivery of a fetus through surgical incisions made through the abdominal wall (laparotomy) and the uterine wall (hysterectomy) Elective cesarean delivery: cesarean delivery is done before the onset of labor when surgeons decided.

NRS: Is a valid pain intensity assessment tool that involves asking a patient to rate his or her pain from 0-10 (11-point scale) with the understanding that 0 is equal to no pain and 10 equal to the worst possible pain Total analgesic consumption: the total amount of analgesic drugs in milligrams used in the first 24 hours after the operation.

Time to first analgesic request: is a time in minutes measured from the end of the procedure to the time when the patient requests analgesics.

Duration of surgery: time in minutes from skin incision to end skin closure. Duration of anesthesia: a time in minutes it takes from administration of induction agent to the time a patient is intubated.

ELIGIBILITY:
Inclusion Criteria:

* Women age between 18 and 35
* ASA risk class I-II

Exclusion Criteria:

* - Chronic pain diagnosis
* ASA above II
* Comorbidities (Anemia, DM, HTN, Arthritis)
* Known allergy to bupivacaine, tramadol
* History of alcohol, opiate, or other drug abuse
* Use of preoperative anti-pain

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The stud focused on a mother giving birth by incision (cesarian section)
Enrollment: 163 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
Measuring pain severity | starting from discharging from operation table to the 2nd day of surgery ( for 48 hours)
  Pain severity is measured by a visual analog scale(VAS) which measures pain severity from zero to ten

CONTACTS AND LOCATIONS:
Overall Officials: Woldemichael, Principal Investigator — Wollo Universty
Locations (1):
- Dessie comprehensive specilized hospital, Dessie, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
we are not sure about sharing until we get the necessary materials but after we get, we are willing to share!